CLINICAL TRIAL: NCT06262282
Title: A Prospective Standardized Assessment of People With Cystic Fibrosis and Non-tuberculosis Mycobacteria Pulmonary Disease Undergoing Treatment With Mycobacteriophage (POSTSTAMP)
Brief Title: Mycobacteriophage Treatment of Non-tuberculosis Mycobacteria
Acronym: POSTSTAMP
Status: Enrolling by invitation | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jerry A. Nick, M.D., Director, Adult Cystic Fibrosis Program, National Jewish Health
Other Study IDs: NTM-OB-17 (PART C)
Record Dates: First submitted 2024-02-04; First posted 2024-02-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis; Nontuberculous Mycobacterial Lung Disease; Nontuberculous Mycobacterium Infection; Mycobacterium Infections; Mycobacterium; Pulmonary
Keywords: cystic fibrosis; phage; mycobacteriophage
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — NTM isolates will be sent to the National Jewish Health (NJH) laboratory for additional testing and will be stored for future research. Specimens will be banked for future research use (blood, sputum, urine, and NTM isolates- including any previous isolates that might be available or previously sent to NJH for analysis). The specimens will be used to learn more about NTM Disease and to learn more about CF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with cystic fibrosis who are receiving phage treatment for NTM.: People with cystic fibrosis who have identified at least one phage effective against their NTM infection and are receiving treatment with the phage. These subjects will remain on guideline based NTM antibiotic treatment and their standard CF care. They will receive therapeutic phage twice daily for 1 year.
  Interventions: Biological: mycobacteriophage
- People with cystic fibrosis who are not receiving phage treatment for NTM.: People with cystic fibrosis who have not identified any phage effective against their NTM infection and are not receiving phage treatment. These subjects will continue with guideline based NTM antibiotic treatment for their NTM disease and standard CF care.

INTERVENTIONS:
Biological: mycobacteriophage — mycobacteriophage phage that has been found effective in killing participants NTM infection
  Groups: People with cystic fibrosis who are receiving phage treatment for NTM.

SUMMARY:
About 10 people with cystic fibrosis (CF) and persistent Nontuberculosis mycobacteria (NTM) infection despite treatment will be screened to find out if their NTM infection has at least one mycobacteriophage that is effective in killing the mycobacteria. Individuals who are found to have at least one phage will be offered assistance in pursuing FDA approval for treatment via expanded-access Individual New Drug (IND) for compassionate-use. They will receive phage treatment for 1 year along with their guideline-based antibiotics for NTM. Individuals who are not identified as having a phage match will be followed as they continue to receive guideline based antibiotic therapy for 1 year. All subjects, including those who do not have a phage match will continue to be observed for the duration of the study, or about 1 year.

DETAILED DESCRIPTION:
About 10 people with cystic fibrosis and NTM infection with positive sputum cultures after a minimum of 12 months of guideline-based therapy will be screened to find out if their NTM infection has at least one mycobacteriophage that is known to be effective against the NTM. Individuals who have been found to have at least one effective phage will be offered assistance in pursuing FDA approval for phage treatment through a compassionate-use Individual New Drug (IND). These subjects will receive phage treatment for 1 year along with their guideline-based antibiotics for NTM. Individuals who are not identified as having a phage match will continue to receive guideline based antibiotic therapy. All subjects, receiving phage or not, will be observed and assessed, including collection of specimens, to evaluate response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative
2. Enrolled in the CFF Patient Registry (CFF PR)
3. Be willing to adhere to study procedures in the context of clinical care, and other protocol requirements
4. Male or female participant ≥ 6 years of age at enrollment who are able to reliably expectorate sputum and/or willing to undergo sputum induction (if necessary)
5. Diagnosis of CF consistent with the 2017 CFF Guidelines
6. NTM pulmonary disease on treatment with guideline-based antibiotics for >12 months without consistent conversion of airway cultures to negative.
7. Physician intention to treat NTM with phage therapy (if susceptible)
8. Be willing and able to continue guideline-based antibiotics for NTM concurrent with phage.
9. Documentation of a sufficient number of NTM cultures with a sufficient proportion of positive cultures in the interval 12 months prior to initiation of phage to allow for a within-subject power ≥0.80 to detect a difference in the percent positive NTM cultures in the interval 6-18 months following initiation of phage.

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Prior or ongoing phage therapy for the species of NTM under consideration.
3. History of solid organ or hematological transplantation
4. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a diagnosis of CF who meet all of the inclusion and none of the exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to therapy | Comparing the year of phage therapy to the year prior to start of phage therapy
  Proportion who adhere to the POSTSTAMP protocol based on number of respiratory cultures obtained per year, withdrawals or major deviations from protocol.

SECONDARY OUTCOMES:
Phage susceptibility | At the time of enrollment
  Proportion of participants with NTM infection susceptible to phage
Culture conversion | Any 12 month interval from the start of phage therapy to end of follow-up, an average of about 2 years.
  Proportion of participants with >12 months of consecutive negative cultures with no subsequent positive cultures.
Tolerance of treatment | From enrollment through study completion, an average of about 24-30 months.
  Proportion requiring antibiotic course change due to intolerance or lack of microbiological conversion (i.e. eradication from sputum)
Clinical Response (pulmonary function testing) | From enrollment through study completion, an average of about 24-30 months.
  Within subject change in forced expiratory volume at one second (FEV1) with increase indicating improvement in lung function or FEV1 decrease indicating decline in lung function.
Microbiologic response to phage | A year interval from month 6 of treatment to month 18 following start of phage will be compared to the year prior to start of phage.
  Within-subject change in percent positive (%pos) cultures following phage initiation (or identification that no phage is available), compared to the interval prior to phage initiation (or identification that no phage is available): the period of antibiotic treatment without phage.
Clinical response (BMI) | From enrollment through study completion, an average of about 24-30 months.
  Within subject change in BMI with decline in BMI as sign of decline or worse outcome.
Clinical response (CFQR) | From enrollment through study completion, an average of about 24-30 months.
  Within subject change in Cystic Fibrosis Questionnaire -Research (CFQR) score, with higher score indicating worse symptoms.
Clinical Response (antibiotic courses for non- NTM exacerbations) | From enrollment through study completion, an average of about 24-30 months.
  Proportion of non-NTM exacerbations compared to NTM exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nick, MD, Principal Investigator — National Jewish Health
Locations (18):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, San Diego, California
  - Childrens Hospital Colorado, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont, Burlington, Vermont
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided